CLINICAL TRIAL: NCT06493981
Title: Long Term Outcomes of Eltrombopag in Patients With Bone Marrow Aplasia, Assiut University Hospital Insight.
Brief Title: Outcomes in Bone Marrow Aplasia.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Mahmoud, Long term outcomes of eltrombopag in patients with bone marrow aplasia, Assiut university hospital insight., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Noha Mahmoud Muhammed
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Aplastic Anemia Idiopathic
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cases of aplastic anemia recieving Eltrombopag (Experimental): Newely diagnosed bone marrow aplasia starting treatment with Eltrombopag in adose of 50-150mg / day
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Treatment with eltrombopag in a dose of (50-150mg/d)
  Other Names: Revolade; Versapenia

SUMMARY:
Bone marrow aplasia, also known as aplastic anemia (AA) is a potentially fatal bone marrow failure syndrome characterized by a paucity of hematopoietic stem cells (HSCs) and progenitor cells with varying degrees of cytopenia and fatty infiltration of the bone marrow space. Underlying mechanisms include immune-mediated attack, telomere defects, and inherent HSC compartment insufficiency. These events may occur individually or in concert, mostly involving effector T cells Historical treatment has included the use of high-dose chemotherapy and allogeneic stem cell transplantation as well as lymphotoxic immunosuppressive therapy (IST) Thrombopoietin (TPO) regulates platelet production, maturation, and release through binding of c-mpl on megakaryocytes.

DETAILED DESCRIPTION:
Eltrombopag (E-PAG) is an oral synthetic small-molecule, noncompetitive, TPO agonist that initially was approved by the US Food and Drug Administration (FDA) for the treatment of chronic immune thrombocytopenic purpura. Single-agent activity of E-PAG was demonstrated in at least 1 lineage in 40 to 45% of patients with AA that was refractory to IST, leading to its approval by the FDA in this setting (5).

Eltrombopag evades cytokines blockade of c-MPL signaling and activates the c-MPL receptor by interacting with the transmembrane receptor domain, resulting in a conformational change without competing with TPO. Regarding AA, it is possible that eltrombopag promotes DNA repair in hematopoietic stem cells and progenitor cells. However, AA may appear to evolve to other hematologic diseases, most notably paroxysmal nocturnal hemoglobinuria and myelodysplastic syndrome, even to acute myeloid leukemia, and about 15% of patients evolve to myelodysplastic syndrome, acute myeloid leukemia or both after immunosuppressive therapy. Therefore, it is unclear but alarming that the use of eltrombopag exacerbates the clone evolution (6).

Eltrombopag and cyclosporin was active as front-line treatment of severe aplastic anaemia, with no unexpected safety concerns. This approach might be beneficial where horse-ATG is not available or not tolerated.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18. Newely diagnosed bone marrow aplasia Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. Patients started CSA plus Eltrombopag therapy Normal cardiac, hepatic & renal functions

Exclusion Criteria:

Hypersensitivity or contraindications to eltrombopag. Cardiovascular, pulmonary, hepatic, or renal diseases. History of malignancy. Pregnant, breastfeeding. Inherited bone marrow aplasia. Secondry bone marrow aplasia Previous thromboembolic events. Previous malignancies either solid or hematologic.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Determine hematological response after 6 months | 6 months to 5 years
  Change in CBC elements after 6 months of treatment
Determine overall survival rate. | 5 years
  Number if years estimated to survive after treatment

SECONDARY OUTCOMES:
Rate of relapse in patients deemed responsers at 6 months. | Around 1 year
Clonal evolution to myeloid malignancy or new chromosomal abnormality | Around 2 years
Change in serum iron and ferritin over time of treatment | From 6 months to 5 years
Eltrombopag efficacy in increasing platelet count | After6 months
Adverse effects raelated to treatment | Within 2 years